CLINICAL TRIAL: NCT02372565
Title: Using Mass Media to Promote Physical Activity in African American Women
Brief Title: Facebook to Promote Physical Activity in Black Women African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Barbara E. Ainsworth, Regents' Professor, Exercise Science and Health Promotion, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000485
Record Dates: First submitted 2015-02-06; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Physical Activity
Keywords: African American; Women; Physical Activity; Social Media; Exercise; Facebook; Text message
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Facebook and Text Message (Experimental): Participants randomized to the technology-based physical activity intervention will receive a culturally-relevant physical activity promotion intervention delivered via text messages and the social media website Facebook. The purpose of the intervention materials is to encourage participants to achieve a minimum of 150 minutes/week of moderate-intensity aerobic physical activity each week.
  Interventions: Behavioral: Facebook and text Message
- Standard Print-based Intervention (Active Comparator): Participants randomized to the standard print-based physical activity intervention group will be mailed 4 self-help booklets promoting physical activity produced by the American Heart Association. Booklets will be mailed one at a time in 2 week intervals over the 1st 6-weeks of the intervention. These high quality booklets provide general information on the benefits of physical activity, tips and strategies to increase daily physical activity, and encourage recipients to perform a minimum of 10,000 steps per day.
  Interventions: Behavioral: Standard Print-based Intervention

INTERVENTIONS:
Behavioral: Facebook and text Message — Culturally-relevant physical activity promotion program
  Arms: Facebook and Text Message
Behavioral: Standard Print-based Intervention — Non-culturally relevant physical activity promotion program
  Arms: Standard Print-based Intervention

SUMMARY:
The purpose of this study is to evaluate the feasibility of a social media and text-message-delivered, Social Cognitive Theory-based, culturally relevant intervention designed to promote physical activity among African American women. An 8-week, 2-arm randomized trial will be implemented. Arm 1 will receive a culturally-relevant, technology-based physical activity intervention delivered via Facebook and text messages. Arm 2 (Comparison Group) will receive a standard print-based physical activity promotion materials consisting of high quality physical activity promotion brochures produced by the American Heart Association.

DETAILED DESCRIPTION:
The purpose of this study is to apply and investigate the feasibility of a social media and text-message-delivered, Social Cognitive Theory-based, culturally relevant intervention designed to promote physical activity among African American women. In an 8-week, 2-arm randomized trial, 30 African American women will be assigned to receive either: a) culturally-relevant, technology-based physical activity intervention delivered via Facebook and text messages, or b) a standard print-based physical activity promotion intervention consisting of high quality physical activity promotion brochures produced by the American Heart Association delivered via USPS mail.

Aim 1: Test the feasibility of a culturally relevant, social media and text-message delivered physical promotion pilot intervention among adult African American women. The investigators hypothesize that the culturally relevant Facebook and text message delivered intervention will be feasible as measured by the acceptability, implementation, and practicality of the intervention program.

Aim 2: Examine the impact of the culturally-relevant, Facebook and text message delivered intervention to increase physical activity and enhance associated Social Cognitive Theory constructs explicitly targeted by the intervention activities. Physical activity will be objectively measured by accelerometers and Social Cognitive Theory constructs of self-efficacy, social support, self-regulation, and outcome expectations will be assessed by validated self-report questionnaires. The investigators hypothesize that participants receiving the culturally-adapted, Social Cognitive Theory-based Facebook and text-message intervention will demonstrate higher physical activity levels and greater enhancements in Social Cognitive Theory constructs when compared to the standard print-based intervention group at the post-intervention assessment.

Aim 3: Examine the preliminary effect of a culturally relevant, social media-delivered physical activity promotion intervention on anthropometric, blood pressure, and blood lipid outcomes. The investigators hypothesize that increased physical activity at the post-intervention follow-up will be associated with improvements in these variables.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as African American
* female
* insufficiently active (<150 min/week of moderate-intensity physical activity assessed by the short version of the International Physical Activity Questionnaire)
* aged 24-49 years
* having an active Facebook account
* ability to read/write in English

Exclusion Criteria:

* concurrent participation in another physical activity promotion program (research or commercial)
* being pregnant or planning on becoming pregnant in the next 6 months, and
* self-reported condition that inhibits engagement in physical activity
* contraindication for physical activity according to the Physical Activity Readiness Questionnaire (PAR-Q) unless written permission from the participant's physician to engage in the study is provided

Ages: 24 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of Using Facebook and Text Messaging to Deliver a Physical Activity Program to African American Women | Post Intervention (up to 8 weeks)
  Measured using a composite score by assessing acceptability (participants perceived satisfaction and usefulness of the program; perceived cultural relevance of the program), demand (interest in study participation; participant retention), and implementation (participant activity on the Facebook group page, successful delivery of text messages, successful delivery of study materials on the study Facebook wall) of the culturally relevant physical activity program.

SECONDARY OUTCOMES:
Change in physical activity from baseline to 8 weeks | Two assessments, 8 weeks apart
  Assessed by ActiGraph GT3X+ accelerometers
Change in exercise self-efficacy from baseline to 8 weeks | Two assessments, 8 weeks apart
  Assessed by the Exercise Confidence Survey (Sallis, 1988)
Change in social support for exercise from baseline to 8 weeks | Two assessments, 8 weeks apart
  Assessed by the Social Support for Exercise Survey (Sallis,1987)
Change in self-regulation for physical activity from baseline to 8 weeks | Two assessments, 8 weeks apart
  Assessed by the Self-Regulation Scale from the Health Beliefs Survey (Anderson, 2010)
Change in outcome expectations for exercise from baseline to 8 weeks | Two assessments, 8 weeks apart
  Assessed by the Outcome Expectation Scale for Exercise (Resnick, 2000)
Change in body mass index (BMI) from baseline to 8 weeks | Two assessments, 8 weeks apart
Change in total serum cholesterol from baseline to 8 weeks | Two assessments, 8 weeks apart
Change in serum high-density lipoprotein (HDL) cholesterol from baseline to 8 weeks | Two assessments, 8 weeks apart
Change in serum low-density lipoprotein (LDL) cholesterol from baseline to 8 weeks | Two assessments, 8 weeks apart
Change in serum triglycerides from baseline to 8 weeks | Two assessments, 8 weeks apart

REFERENCES:
- [Derived] Joseph RP, Keller C, Adams MA, Ainsworth BE. Print versus a culturally-relevant Facebook and text message delivered intervention to promote physical activity in African American women: a randomized pilot trial. BMC Womens Health. 2015 Mar 27;15:30. doi: 10.1186/s12905-015-0186-1. PMID 25886945